CLINICAL TRIAL: NCT06418516
Title: Early Detection of Esophageal Squamous Cell Carcinoma With the Capsule Sponge Device Coupled With Molecular Biomarkers and Machine Learning
Brief Title: Early Detection of Esophageal Squamous Cancer With the Capsule Sponge Device
Acronym: ANGELA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Collaborators: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 439/2023
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Cancer; Head and Neck Cancer; Squamous Cell Carcinoma
Keywords: Prevention; Screening; Esophageal Cancer; Capsule Sponge
MeSH Terms: conditions — Esophageal Neoplasms; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Gastroscopy; Biopsy; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Single Group Assignment A prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Capsule-sponge (Experimental): This part of the study will have an active prospective recruitment of patients. Recruitment will involve three patient populations:
  1. Patients with ESCC
  2. Patients at high risk for ESCC
  3. Healthy controls
  Following inclusion in the study, subjects will be asked to complete a behavior questionnaire, have blood collected, and undergo a capsule-sponge procedure followed by diagnostic gastroscopy using advanced imaging with biopsies. During gastroscopy, additional tissue samples will be collected for research purposes. These samples, along with cytological specimens from the capsule-sponge, will be analyzed to assess the diagnostic accuracy of biomarkers in the diagnosis of esophageal squamous neoplasia.
  Interventions: Device: Capsule-sponge

INTERVENTIONS:
Device: Capsule-sponge — The capsule-sponge is a minimally-invasive sampling device consisting of a polyurethane sponge compressed in a cellophane capsule attached to a string. When swallowed, the capsule dissolves in the stomach, releasing the cell collection sponge that expands to 3 cm in diameter. Next, a nurse or qualified medical technician retrieves the sponge by pulling back on the string and retracting it through the mouth. During extraction, the rough texture on the surface of the sponge collects epithelial cells in the cardia and along the entire length of the esophagus.
  Other Names: Upper endoscopy with biopsies; Blood collection; throat swab

SUMMARY:
Esophageal squamous cell carcinoma accounts for ~90% of the nearly half-million annual incident cases of esophageal cancer worldwide. The high costs and invasiveness of upper endoscopy constitute a limitation in providing adequate surveillance for at-risk individuals, including those with previous head and neck cancer. The ANGELA study is a prospective evaluation of the minimally-invasive capsule-sponge device, coupled with tissue biomarkers (p53-immunohistochemistry), to detect squamous neoplasia in high-risk individuals.

DETAILED DESCRIPTION:
Esophageal squamous cell carcinoma (ESCC) is the most common type of esophageal cancer worldwide, accounting for nearly 90% of the 456,000 incident cases of esophageal cancer each year. Overall, it is the seventh most common malignancy and the sixth most common cause of cancer-related mortality, with a high incidence rate in eastern to central Asia and eastern and southern Africa. This cancer is more common in men (~70%), and the main risk factors include cigarette smoking, alcohol consumption, poor oral hygiene, the ingestion of caustic agents, and nutritional deficiencies. Additionally, an increased risk of ESCC following curative treatment of head and neck cancer (HNC) has been well-documented in the literature, with a lifetime incidence ranging between 3.8% and 14.9% in prospective observational studies. The carcinogenesis of ESCC is sequential and preceded by several precancerous stages, including low-grade intraepithelial neoplasia (LG-IEN) and, subsequently, high-grade intraepithelial neoplasia (HG-IEN).

Although the prognosis of ESCC is extremely poor, with 5-year survival below 20%, it dramatically improves if the disease is detected at an early stage. Consequently, mass screening in high-incidence regions is being widely debated. However, population-wide screening presents a large challenge in terms of cost-effectiveness and manpower, as currently, a potential screening regime for ESCC would rely on endoscopic examination with biopsies, which remains the gold standard for ESCC diagnosis. Furthermore, since around 80% of all ESCCs occur in economically less-developed regions, newer, cheaper, and less invasive diagnostic tools are highly warranted.

The capsule-sponge is a novel, minimally-invasive device that collects cells from the esophagus to produce a pseudo-biopsy suitable for routine laboratory analysis. In addition, tissue biomarkers such as p53 immunohistochemistry (p53-IHC) and molecular testing, including copy number assays to detect aneuploidy, can be applied. There is extensive data on the use of this technology for early diagnosis of Barrett's esophagus (precursor to adenocarcinoma), which has now reached wide clinical implementation in the UK National Health Service. Building on the promising pilot data, the current study aims to expand further our previously developed clinical assay for early detection of esophageal squamous neoplasia using the capsule-sponge device coupled with biomarkers and machine learning technologies.

In this prospective trial, we plan to recruit patients within three risk groups for ESCC: 1. healthy controls; 2. high-risk individuals (previous head-and-neck cancer/ESCC); and 3. patients with known early ESCC. Each patient will undergo a high-definition endoscopy and a capsule-sponge examination. The biomarker assay, including p53-IHC and shallow whole genome sequencing, will be tested within the capsule-sponge samples and compared with the final endoscopic diagnosis. Machine learning algorithms will be applied to digitalized cytology to detect atypical cells and regions of p53-IHC overexpression. Lastly, we will extract microbial DNA from capsule-sponge samples to assess any taxonomic diversity within the three risk groups for ESCC.

We hope to develop a novel, effective, and affordable diagnostic assay that, coupled with a minimally-invasive capsule-sponge device, could be implemented in a clinical setting, improving the early detection of ESCC and, eventually, patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with esophageal squamous cell cancer (ESCC):

   * Patients ≥18 years of with adequate performance status for endoscopy
   * Newly diagnosed ESCC suitable for endoscopic or oncological treatment (Rth/Chth)
   * Patients currently undergoing oncological treatment (Rth/Chth)
   * Consent to provide tissue samples for the study
   * Dysphagia grade ≤2 (able to swallow mixed foods and tablets)
2. Patients at high risk for ESCC:

   * Patients ≥18 years of age with adequate performance status for endoscopy
   * Prior definitive treatment for head and neck cancer (cancer of the oral cavity, hypopharyngeal cancer, laryngeal carcinoma) and at least 12 months post-therapy (both Rth, Chth, and combination treatment)
   * Prior definitive endoscopic treatment for early ESCC in the past (at least 6 months since completion)
   * Consent to provide tissue samples for the study
   * Dysphagia grade ≤2
3. Healthy controls - Patients ≥18 years old undergoing endoscopic evaluation for typical GI symptoms other than dysphagia (e.g., GERD, dyspepsia, etc.) without significant risk factors for ESCC

Exclusion Criteria (for all patients):

* Patients currently on anticoagulant treatment (warfarin, acenocoumarol) with no possibility of stopping / modification
* Dysphagia grade ≥3 (able to swallow only liquid foods)
* History of myocardial infarction or other cardiovascular event within 6 months of enrolment
* Neurological diseases associated with impaired swallowing
* Patients in long-term care or institutional care (physical, psycho-social disorders, intellectual disability).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility and diagnostic yield of capsule-sponge coupled with cellular atypia and p53-IHC analysis for detecting ESCC and its precursor lesions compared with endoscopy (gold standard) | 3 years
  Sensitivity (%) and Specificity (%) of the capsule-sponge device in identifying patients with early squamous neoplasia (LG-IEN, HG-IEN, ESCC) as compared to the upper endoscopy with biopsies (gold standard)

SECONDARY OUTCOMES:
Acceptability of the capsule-sponge device in patients with ESCC and high-risk for ESCC | 3 years
  % of Participants that have scored the Cytosponge experience of at least 6 points on a 0 to 10 Visual Analogue Scale (VAS) acceptability scale whereby 0 denotes "worst experience in life" and 10 denotes "best experience in life".
Study on accuracy and feasibility of adding copy number profiling for aneuploidy assessment to the capsule-sponge samples | 3 years
  Within this outcome, we will clarify the optimal depth of sequencing, and we will then perform shallow whole genome sequencing (sWGS) on the samples collected in the training phase to input the copy-number variation (CNV) into the classification algorithm and evaluate the output as compared with the diagnosis of the patient. This will enable us to refine the classifications with the ultimate aim of using them predictively in a testing phase.
Application of artificial intelligence on Cytosponge digitalized samples | 3 years
  To assess the utility of machine learning-based approaches to assist pathological assessment of the capsule-sponge samples for the applicability of the technology at scale. We will test the feasibility of applying the artificial intelligence (AI)-based technology onto digitalized capsule-sponge samples. The assessment will comprise of AI training phase and a validation period.

CONTACTS AND LOCATIONS:
Overall Officials: Wladyslaw Januszewicz, M.D., PhD, Principal Investigator — Centre of Postgraduate Medical Education, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Data obtained through this study may be provided to qualified researchers with academic interest in esophageal cancer. Data or samples shared will be coded. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.